CLINICAL TRIAL: NCT04516876
Title: Efficacy Research of Bimanual Intensive Training in Children With Hemiplegic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202004060RIND
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy, bimanual intensive training, occupational therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camp-based bimanual intensive training(BIT) (Experimental)
  Interventions: Other: Camp-based bimanual intensive training(BIT)

INTERVENTIONS:
Other: Camp-based bimanual intensive training(BIT) — The day-camp BIT model will be delivered in a group-based design. In day-camp model, each child is assigned to a trained therapist to maintain at least a 1:1 to 1:2 ratios of therapy and child. The therapist will monitor and modify the activities to fit each individual's ability and need to make sure the intervention quality is equivalence to the individualized treatment method. The chosen tasks of each intervention session have to be considering the child's preference, age-appropriated, and at the right level of difficulty. Target movements are embedded in the functional activities, whereby the environment is manipulated to vary task requirement and the difficulty is graded to match the child's capacity.

SUMMARY:
This research project aims to investigate the feasibility, efficacy, and acceptability of camp-based model of BIT.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cerebral palsy(CP) with one or more affected sides.
2. Considerable nonuse of the affected upper limb (amount-of-use score of the Pediatric Motor Activity Log < 2.5).
3. No excessive muscle tone (Modified Ashworth Scale ≤ 2 at any joints of the upper limb) before beginning treatment.
4. No severe cognitive, visual, or auditory disorders according to medical documents, parental reports, and the examiner 's clinical observation.
5. No injections of botulinum toxin type A or operations on the upper limb within 6 months.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-08-03 (Estimated); Study Completion 2024-08-03 (Estimated)

PRIMARY OUTCOMES:
Score changes of Melbourne Assessment 2 | baseline, after one week, after 2 months, after 6 months
  The Melbourne Assessment 2(MA2) was developed to investigate the objective upper-limb movement in children with CP aged 2.5 to 15 years.The four main elements of movement quality include (1) amount of active ROM; (2) accuracy; (3) dexterity of finger movements; and (4) fluency or smoothness of movement. The scoring sheet consists of 3-, 4-, or 5-point scales from 0 to 4 that allocate scores on the 14 items.Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Score changes of Bruininks-Oseretsky Test of Motor Proficiency | baseline, after one week, after 2 months, after 6 months
  The subtest 3 of the Bruininks-Oseretsky Test(BOT-2), manual dexterity (MD), will be used to assess a child's upper limb dexterity. The subtests 3 of the BOT-2 consist of 5 goal-directed activities that involve reaching, grasping, and bimanual coordination with small objects to investigate a child's upper limb manual function.Higher scores mean a better outcome.
Score changes of Box and Block test | baseline, after one week, after 2 months, after 6 months
  The Box and Block test (BBT) assesses manual dexterity by county the number of blocks that are transferred with a single hand from one compartment to another within 60 seconds.Higher scores mean a better outcome.
Performance changes of motion analysis | baseline, after one week, after 2 months, after 6 months
  Three-dimensional marker trajectory data will be measured using a motion analysis system (Vicon MX, Oxford Metrics Group, U.K.). Twenty-eight passive infrared retroreflective markers will be attached to the skin of the body segments to track the motion of the body segments. For the performance outcome measures, endpoint variables during reach-to-grasp task, namely reaction time, movement time, movement unit, peak velocity and its time percentage during the movement time will be calculated using the wrist marker. For the performance production measures, joint angles of the shoulder, elbow and wrist during reach-to-grasp task will also be calculated to represent the motor strategy of children with CP before and after intervention.
Score changes of Pediatric Motor Activity Log-Revised | baseline, after one week, after 2 months, after 6 months
  The Pediatric Motor Activity Log-Revised(PMAL-R) is a parent-reported evaluative tool used to capture the spontaneous use of the affected upper limb in 22 daily activities. Each activity is rated by parents/careers on two set (how often and how well) of 6-point ordinal scales (0-5). The 'how often' scale measures amount of use, and the 'how well' scale measures quality of movement, of the affected upper limb.Higher scores mean a better outcome.
Score changes of ABILHAND-kids Questionnaire | baseline, after one week, after 2 months, after 6 months
  The ABILHAND-Kids questionnaire is a Rasch-based assessment that measures children's perceived difficulty in performing ADL that require the use of the bilateral upper limbs. It contains 21 items measuring manual ability and is rated on a 3-point response scale(0-2). The parent is asked to fill in the questionnaire by estimating their child's ease or difficulty in performing each activity, irrespective of the limb(s) the child actually use and whatever the strategies used to perform the activity.Higher scores mean a better outcome .
Score changes of Pediatric Evaluation of Disability Inventory | baseline, after one week, after 2 months, after 6 months
  The Pediatric Evaluation of Disability Inventory(PEDI) is a parent-reported questionnaire. It contains two subscales :(1)functional skill scale (2)caregiver assistance scale. The parent is asked to fill in the questionnaire by estimating their child's performance capability in 197 items in three domains :(1)self-care (2)mobility (3)social is rated on a 2-point response scale(0-1). In caregiver assistance scale, the needs of caregiver assistance to complete each activity are scored from 0 to 5 point.Higher scores mean a better outcome in both parts .
Score changes of Dimensions of Mastery Questionnaire | baseline, after one week, after 2 months, after 6 months
Score changes of Test of Playfulness | from the first day to the sixth day of the intervention
Score changes of Pediatric Engagement Questionnaire | from the first day to the sixth day of the intervention
Score changes of Client Satisfaction Questionnaire | from the first day to the sixth day of the intervention
Score changes of Parenting Stress Index-Short Form | baseline, after one week, after 2 months, after 6 months
  The Parenting Stress Index-Short Form(PSI-SF) is direct derivative from the Parenting Stress Index (PSI) full-length test which was created to sample a diverse range of potential influences on parenting practices to address the need for a psychometrically sound but brief screening measure of parenting stress. All 36 items of the PSI-SF consist of three subscales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. Each subscale consists of 12 items rated from 1 (strongly disagree) to 5 (strongly agree). High scores on the subscale and PSI-SF total score indicate greater level of stress

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Department of Occupational Therapy, Taipei, Taiwan